CLINICAL TRIAL: NCT05323708
Title: A Randomized, Double-blind, Two-arm, Single-dose, Parallel-Group Study to Compare the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Bmab 1000 and Prolia® in Normal Healthy Volunteers
Brief Title: Comparison of Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Bmab 1000 and Prolia® in Normal Healthy Volunteers: DENARIUS: DENosumab Pharmacokinetic equivAlence tRIal in Healthy volUnteerS
Acronym: DENARIUS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocon Biologics UK Ltd (Industry)
Collaborators: Biotrial (Industry)
Responsible Party: Sponsor
Organization: Biocon Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1000-NHV-01-G-01
Record Dates: First submitted 2022-03-15; First posted 2022-04-12 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind (Patient, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bmab 1000, A single 60 mg dose of Bmab 1000 administered by subcutaneous injection. (Experimental)
  Interventions: Biological: Bmab 1000
- Prolia®, A single 60 mg dose of Prolia® administered by subcutaneous injection. (Active Comparator)
  Interventions: Biological: Prolia®

INTERVENTIONS:
Biological: Bmab 1000 — 60mg/ml Prefilled syringe single dose
  Arms: Bmab 1000, A single 60 mg dose of Bmab 1000 administered by subcutaneous injection.
Biological: Prolia® — 60mg/ml Prefilled syringe single dose
  Arms: Prolia®, A single 60 mg dose of Prolia® administered by subcutaneous injection.

SUMMARY:
This study is to compare the Pharmacokinetics, Pharmacodynamics, safety, and tolerability of Bmab 1000 and Prolia® in normal healthy volunteers.

DETAILED DESCRIPTION:
This study will consist of 2 study periods: Screening period (4 weeks) and Treatment period (Dosing and follow-up).

In this double-blind, 2-arm study, the eligible subjects will be randomized in a 1:1 ratio to receive either Bmab 1000 or Prolia® on Day 1. The interventions (Bmab 1000 or Prolia®) will be administered subcutaneously. End-of-study visit will be at Week 36 post randomization.

The total duration of study participation for a subject will be up to 40 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: Male or Female
2. Age: Male subjects: 28-55 years, inclusive at screening; Female subjects: 28-45 years, inclusive at screening.
3. Weight: For non-Japanese subjects 60.0-95.0 kg, inclusive at screening. For Japanese subjects 55.0-95.0 kg, inclusive at screening.
4. Body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive, at screening.
5. Vital signs showing no clinically relevant deviations according to the Investigator's judgment or their designee's. In the case of subjects > 45 year-old, if a value of SBP above 145 mmHg is confirmed on rechecking the BP after a period of rest, this subject will not be included in the study.
6. 12-lead ECG recording without signs of clinically relevant pathology or showing no clinically relevant deviations as judged by the Investigator or their designee.

Exclusion Criteria:

1. Evidence of clinically relevant pathology: Like have a history of and/or current clinically significant gastrointestinal, renal, hepatic, cardiovascular, haematological, pulmonary, neurologic, metabolic, psychiatric disorder, drug or alcohol abuse, or allergic disease excluding mild asymptomatic seasonal allergies. Have a history of malignancy (including lymphoma, leukaemia, and skin cancer).
2. Unable to follow protocol instructions or not likely to complete the study in the opinion of the Investigator or their designee.
3. History of relevant drug and/or food allergies (including hypersensitivity to any recombinant protein drug or any of the constituents of denosumab, or latex allergy or hereditary problems of fructose intolerance).
4. Known history of previous exposure to denosumab.
5. Have previously been exposed to a monoclonal antibody or fusion protein (other than denosumab) within 270 days (or 5 half-lives whichever is the longest) prior to randomization and/or there is confirmed evidence or clinical suspicion of immunogenicity from previous exposure to a monoclonal antibody or fusion protein.
6. Prior diagnosis of bone disease, or any condition that will affect bone metabolism such as, but not limited to: osteoporosis, osteogenesis imperfect, hyperparathyroidism, hyperthyroidism, hypothyroidism, osteomalacia, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, current flare-up of osteoarthritis and/or gout, active malignancy, renal disease (defined as glomerular filtration rate < 60 mL/min), Paget's disease of the bone, recent bone fracture (within 6 months), malabsorption syndrome.
7. Any use of the following bone modifying medications, with no limitation on time since administration: e.g.intravenous bisphosphonates, strontium, fluoride (if administered in treatment of osteoporosis),romosozumab, teriparatide or any parathyroid hormone analogs, calcitonin, and cinacalcet.

Ages: 28 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
AUCinf (Area Under the Concentration infinity) | 0 to 36 week
  Area under the concentration-time curve from time zero to infinity
AUClast (Area Under the Concentration last) | 0 to 36 week
  Area under the concentration-time curve from time zero to last quantifiable concentration
Cmax | 0 to 36 week
  Maximum serum concentration

SECONDARY OUTCOMES:
Tmax | 0 to 36 week
  Time to reach Cmax
t1/2 | 0 to 36 week
  Terminal half-life
Kel | 0 to 36 week
  Terminal elimination rate constant (kel)
Vd/F | 0 to 36 week
  Apparent volume of distribution
Cl/F | 0 to 36 week
  Apparent clearance
AUEC of sCTX | 0 to 36 week
  Area under the effect curve (AUEC) of serum concentration of C-terminal telopeptide of Type 1 collagen (sCTX)
Emax of sCTX | 0 to 36 week
  Maximal inhibitory effect (Emax) of sCTX
Incidence of TEAEs(Treatment Emergent Adverse Events) | 0 to 36 week
  Experience at least 1 TEAE
Incidence of SAEs(Serious Adverse Events) | 0 to 36 week
  Experience at least 1 SAE
Incidence of ADAs (Anti-Drug Antibodies) | 0 to 36 week
  Incidence of ADAs to denosumab
Titer of ADAs | 0 to 36 week
  Titer of ADAs to denosumab

CONTACTS AND LOCATIONS:
Locations (1):
- Biotrial Inc, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No